CLINICAL TRIAL: NCT00564226
Title: A Placebo Controlled Randomized, 12-week, Dose-ranging, Double-blind Study Versus Placebo Using Tolterodine as a Study Calibrator, to Evaluate Efficacy and Safety of SSR240600C in Women With Overactive Bladder Including Urge Urinary Incontinence
Brief Title: SSR240600C Treatment in Women With Overactive Bladder
Acronym: BILADY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6271; EudraCT 2007-004126-24
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Overactive Bladder
Keywords: urge urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SSR240600C Dose Level 1 (Experimental)
  Interventions: Drug: SSR240600C
- SSR240600C Dose Level 2 (Experimental)
  Interventions: Drug: SSR240600C
- SSR240600C Dose Level 3 (Experimental): dose level 3
  Interventions: Drug: SSR240600C
- Tolterodine (Active Comparator)
  Interventions: Drug: tolterodine
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SSR240600C — oral administration
  Arms: SSR240600C Dose Level 1; SSR240600C Dose Level 2; SSR240600C Dose Level 3
Drug: tolterodine — oral administration
  Arms: Tolterodine
Drug: placebo — oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of SSR240600C in women with overactive bladder compared to placebo using tolterodine as a study calibrator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder

Exclusion Criteria:

* Stress incontinence or mixed incontinence where stress incontinence is the predominant component based on prior history
* Urinary incontinence due to cause other than detrusor overactivity (eg, overflow incontinence)
* Current Urinary Tract Infection (UTI) or frequent UTIs
* Urinary retention or other evidence of poor detrusor function
* Pain during voiding or bladder pain without voiding
* History of radiation cystitis or history of pelvic irradiation
* History of interstitial cystitis or bladder related pain syndrome

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of micturitions per 24 hours | at week 12

SECONDARY OUTCOMES:
Changes from baseline in number of urge urinary incontinence episodes, in number of urgency episodes, in number of nocturia episodes, in volume of urine per void | at week 12
Safety of SSR240600C | at week 12
Quality of life | at week 12

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Aministrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal